CLINICAL TRIAL: NCT01468402
Title: Predictive Factors of Pelvic Magnetic Resonance in the Response of Arterial Embolization of Uterine Leiomyoma
Status: Completed | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Eduardo Zlotnik, Principal Investigator, Hospital Israelita Albert Einstein
Other Study IDs: HIAE
Record Dates: First submitted 2011-10-23; First posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Exposure to Magnetic Field; Uterine Leiomyoma
Keywords: Leiomyoma; uterine artery embolization; magnetic resonance imaging
MeSH Terms: conditions — Myofibroma; Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Magnetic Resonanse Image: The leiomyomas were evaluated individually. MR was used to evaluate morphology: the radiological dimension(s) of the leiomyoma and uterus and the volume. The number of leiomyoma fibroid, and their location in the myometrium was classified. Perfusion and the characterization of the T2 signal were also evaluated.
  Interventions: Procedure: Magnetic Resonance Image

INTERVENTIONS:
Procedure: Magnetic Resonance Image — The leiomyomas were evaluated individually. MR was used to evaluate morphology: the radiological dimension(s) of the leiomyoma and uterus and the volume. The number of leiomyoma fibroids was determined, and their location in the myometrium. Perfusion and the characterization of the T2 signal were also evaluated.
  Other Names: Magnetic Resonance Image with a high-field scanner; Siemens Magnetom 3-Tesla

SUMMARY:
The purpose of this study is to determine predictive factors in the pelvic magnetic resonance in the response of arterial embolization of uterine leiomyoma.

DETAILED DESCRIPTION:
This study followed symptomatic premenopausal women with uterine leiomyoma who underwent uterine artery embolization (UAE). Treatment was accompanied by magnetic resonance imaging of both the volume of the entire uterus and the leiomyomas one month before and six months after UAE. This patients were treated at the Uterine Leiomyoma Sector of the Department of Obstetrics and Gynecology, Medicine College of the University of São Paulo. In this study, the investigators examined 179 leiomyomas in 50 patients.

ELIGIBILITY:
Inclusion Criteria:

* ultrasound diagnosis of uterine leiomyoma
* presence of symptoms (menorrhalgia and/or pelvic pain)
* indication for UAE(the desire to keep the uterus and/or contraindications for surgery).

Exclusion Criteria:

* malignant genital neoplasms
* pelvic inflammatory disease
* allergy to iodinated contrast
* coagulopathy, renal failure
* vasculitis
* pelvic irradiation
* pregnancy
* subserosal leiomyoma with a pedicle smaller than 50% of diameter of the fibroid.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women from the Leiomyoma Service, with eligible criteria and chose this kind of treatment between september 2008 and march 2009.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-09; Primary Completion 2009-04 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Leiomyoma reduction in patients who underwent uterine artery embolization | One month before(baseline) and six month after the embolization
  Use the magnetic resonanse to evaluate factors that predicted leiomyoma reduction in patients who underwent uterine artery embolization

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Zlotnik, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Affonso BB, Nasser F, de Jesus Silva SG, Silva MC, Zlotnik E, de Lorenzo Messina M, Baracat EC. [Strategies for reduction of exposure to ionizing radiation in women undergone to uterine fibroid embolization]. Rev Bras Ginecol Obstet. 2010 Feb;32(2):77-81. Portuguese. PMID 20305945
- [Background] Nasser F, Affonso BB, de Jesus-Silva SG, Coelho Dde O, Zlotnik E, Messina Mde L, Baracat EC. [Uterine fibroid embolization in women with giant fibroids]. Rev Bras Ginecol Obstet. 2010 Nov;32(11):530-5. doi: 10.1590/s0100-72032010001100003. Portuguese. PMID 21271163